CLINICAL TRIAL: NCT01631864
Title: A Randomized, Double-blind, Parallel Group Study to Evaluate Metabolic Effects of LCZ696 and Amlodipine in Obese Hypertensive Subjects
Brief Title: Evaluation of the Metabolic Effects of LCZ696 and Amlodipine in Obese Hypertensive Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: CLCZ696B2207; 2012-002606-40 (EudraCT Number)
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-06

CONDITIONS: Hypertension; Concurrent Obesity
Keywords: Hypertension, obesity, insulin sensitivity, lipolysis, LCZ696
MeSH Terms: conditions — Hypertension; Obesity; Insulin Resistance | interventions — sacubitril and valsartan sodium hydrate drug combination; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCZ696 (Experimental): LCZ696 400 mg plus placebo to amlodipine once daily for 8 weeks
  Interventions: Drug: LCZ696; Drug: Placebo
- amlodipine (Active Comparator): amlodipine 10 mg plus placebo to LCZ696 once daily for 8 weeks
  Interventions: Drug: amlodipine; Drug: Placebo

INTERVENTIONS:
Drug: LCZ696 — LCZ696 was provided as 400 mg tablets.
  Arms: LCZ696
Drug: amlodipine — amlodipine was provided as 5 mg tablets.
  Arms: amlodipine
Drug: Placebo — Matching placebo to LCZ696 and amlodipine.

SUMMARY:
This study investigated the effects of LCZ696 on insulin sensitivity, lipolysis, and oxidative metabolism in obese hypertensive subjects.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any study assessment is performed.
* Males and females of non-childbearing potential ≥ 18 years of age.
* Subjects with mild to moderate essential hypertension,

  * Untreated subjects must have a mean seated SBP (msSBP) ≥ 130 mmHg and < 180 mmHg at screening.
  * Pre-treated subjects must have a msSBP ≤ 160 mmHg at screening and < 180 mmHg at the end of the washout period.
* Waist circumference ≥ 102 cm (men) and ≥ 88 cm (women);

Exclusion criteria:

* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer; or longer if required by local regulations.
* History of angioedema, drug-related or otherwise
* History of hypersensitivity to LCZ696, amlodipine, or drugs of similar chemical classes.
* Severe hypertension (grade 3 of WHO classification; msDBP ≥100 mmHg and/or msSBP ≥ 180 mmHg) at screening or at the end of the washout period.
* Type 1 or Type 2 diabetes mellitus.
* Dyslipidemia requiring pharmacological therapy with a fibrate or nicotinic acid.
* Concomitant use of anti-hypertensives, anti-diabetics, or drugs with effects on glucose or lipid metabolism for the duration of the study.

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Germany (2):
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Neuss
- Novartis Investigative Site, Maastricht, Netherlands

REFERENCES:
- [Derived] Engeli S, Stinkens R, Heise T, May M, Goossens GH, Blaak EE, Havekes B, Jax T, Albrecht D, Pal P, Tegtbur U, Haufe S, Langenickel TH, Jordan J. Effect of Sacubitril/Valsartan on Exercise-Induced Lipid Metabolism in Patients With Obesity and Hypertension. Hypertension. 2018 Jan;71(1):70-77. doi: 10.1161/HYPERTENSIONAHA.117.10224. Epub 2017 Nov 27. PMID 29180454

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCZ696 | Amlodipine
Started | 50 | 48
Completed | 48 | 44
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 | Amlodipine | Total
Number analyzed (Participants) | 50 | 48 | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (9.6) | 50.5 (9.4) | 51.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 41 | 35 | 76

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Insulin Sensitivity Index
Description: The insulin sensitivity index was assessed by hyperinsulinemic euglycemic clamp (HEGC). A positive change from baseline indicates improvement.
Time Frame: baseline, 8 weeks
Population: Pharmacodynamic Analysis Set (PDS): Only participants from the PDS, who had both baseline and day 56 values, were included in the analysis. The PDS included all randomized participants who received at least one dose of study drug and had no protocol deviations with relevant impact on PD data.
Measure: Mean (95% Confidence Interval); unit: ug/kg*min/(mmol/L*pmol/L)
Arm/Group | LCZ696 | Amlodipine
Number analyzed (Participants) | 48 | 41
ug/kg*min/(mmol/L*pmol/L) | 0.192 [0.025 to 0.359] | 0.065 [-0.0116 to 0.246]

2. Secondary Outcome: Local Adipose Tissue Lipolysis, Glycerol Concentrations
Description: Lipolysis was assessed through subcutaneous adipose tissue microdialysis. The actual measure type is adjusted geometric mean.
Time Frame: 57 days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: micro mol/L
Arm/Group | LCZ696 | Amlodipine
Number analyzed (Participants) | 47 | 42
micro mol/L | 82.46 [74.53 to 91.23] | 65.91 [59.22 to 73.37]

3. Secondary Outcome: Oxidative Metabolism
Description: Oxidative metabolism was assessed by indirect calorimetry.
Time Frame: 57 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: carbon dioxide to oxygen ratio
Arm/Group | LCZ696 | Amlodipine
Number analyzed (Participants) | 46 | 40
carbon dioxide to oxygen ratio | 0.787 [0.760 to 0.814] | 0.775 [0.746 to 0.804]

4. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Deaths
Description: Adverse event monitoring was conducted throughout the study.
Time Frame: 8 weeks
Population: Safety Analysis Set (SAS): The SAS included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | LCZ696 | Amlodipine
Number analyzed (Participants) | 50 | 48
Participants
  Adverse events (serious and non-serious) | 30 | 37
  Serious adverse events | 1 | 1
  Deaths | 0 | 0

ADVERSE EVENTS:
Arm/Group | LCZ696 | Amlodipine
Serious Adverse Events (participants affected / at risk) | 1/50 | 1/48
Other Adverse Events (participants affected / at risk) | 23/50 | 26/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=50) | Amlodipine (N=48)
RUPTURED CEREBRAL ANEURYSM (Nervous system disorders) | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=50) | Amlodipine (N=48)
DIARRHOEA (Gastrointestinal disorders) | 3 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 16
NASOPHARYNGITIS (Infections and infestations) | 9 | 8
DIZZINESS (Nervous system disorders) | 3 | 1
HEADACHE (Nervous system disorders) | 4 | 6
PRURITUS (Skin and subcutaneous tissue disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.